CLINICAL TRIAL: NCT00581672
Title: Anxiety in Black Men With Prostate Cancer: Validation of the Memorial Anxiety Scale for Prostate Cancer in an Sample of Black Men
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University School of Medicine(VA-NYU) (Unknown); State University of New York - Downstate Medical Center (Other); Kings County Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-125; NCT00602654 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: Anxiety; Black men; Prostate Cancer; 07-125
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- questionnaires: Black men with prostate cancer
  Interventions: Behavioral: questionnaires of quality of life

INTERVENTIONS:
Behavioral: questionnaires of quality of life — Subjects will be asked to complete the MAX-PC along with additional psychosocial questionnaires which include anxiety, depression coping methods, resilience spirituality, religiosity, and quality of life measures and will take approximately one 30 to 45 minutes to complete by patient.

SUMMARY:
This study is being done to see if a standard tool used to check anxiety in white men works well for Black men. The tool is used only for men who have prostate cancer. It is meant to see how the cancer affects men. If the investigators have a good tool, it is more likely that the investigators can help those who have high levels of anxiety. This test is known as the Memorial Anxiety Scale for Prostate Cancer (also called the MAX-PC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients who are being monitored by PSA tests, who will have a PSA test done on the day of their current clinic visit or prior to their clinic visit, but prior to being informed of the results
* Diagnosis of prostate cancer
* Ethnicity: Black, African-American, or of African descent (and will include those men who identify as Black and Hispanic).
* Ability to comprehend and complete questionnaires in English

Exclusion Criteria:

* Major psychopathology or cognitive impairment likely, in the judgment of the research staff, to interfere with the participation or completion of the protocol
* Other non-Black or non-African-American ethnic groups

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Black men with prostate cancer
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-07-25 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
To establish the psychometric properties of the Memorial Anxiety Scale for Prostate Cancer (MAX-PC) in Black men with prostate cancer. | within one to three weeks of receiving their PSA scores from their physician

SECONDARY OUTCOMES:
To explore the prevalence of distress, anxiety, and depression in Black men with prostate cancer. | within one to three weeks of receiving their PSA scores from their physician

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Downstate Medical Center, Brooklyn, New York
  - Kings County Hopsital Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Martin CM, Schofield E, Napolitano S, Avildsen IK, Emanu JC, Tutino R, Roth AJ, Nelson CJ. African-centered coping, resilience, and psychological distress in Black prostate cancer patients. Psychooncology. 2022 Apr;31(4):622-630. doi: 10.1002/pon.5847. Epub 2021 Nov 9. PMID 34751457
- See also: Memorial Sloan Kettering Web Site — http://www.mskcc.org